CLINICAL TRIAL: NCT06261775
Title: Effect of Minimally Processed Animal Protein on Biomarkers for Cognitive Decline
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Dakota State University (Other)
Responsible Party: Principal Investigator, Moul Dey, Professor, South Dakota State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB-2401011-EXM
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Healthy Lifestyle

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Low UPF no meat
  Interventions: Other: Red meat-based meal; Other: No meat diet
- Test (Experimental): Low UPF with Red meat
  Interventions: Other: Red meat-based meal; Other: No meat diet

INTERVENTIONS:
Other: Red meat-based meal — Participants were provided with food as part of a meal plan. The research team provided all foods and snacks for the intervention.
Other: No meat diet — Participants were provided with food as part of a meal plan. The research team provided all foods and snacks for the intervention.

SUMMARY:
Minimally processed animal protein is a premier source of essential macro and micronutrients in the diet and is important, especially to older adults who are at increased risk of nutritional deficiency and age-related physiological changes. Our central hypothesis is that adding lean animal protein within a healthy diet following macronutrient recommendations for Americans will enhance nutrient adequacy and attenuate markers of cognitive decline. This is a retrospective study leveraging samples collected from the feeding trial NCT05581953. PI for both studies are the same.

ELIGIBILITY:
Inclusion Criteria:

* Generally, good health status based on one routine physical in the past 15 months, current health status
* Normal HbA1C, weigh 110 lb or more
* Age 65 years or more, generally healthy, all races and both sexes
* Generally practicing a meat-based dietary pattern, do not have any special dietary requirements, and
* Willingness to comply with the study protocol, including on-site meal consumption and sample/data collection.

Exclusion Criteria:

* Medication usage, probiotic, long-term antibiotic, and tobacco/drug/alcohol use
* Not on any special diet within 3 months of recruitment, and do not intend to lose weight
* Impaired kidney functions
* Active history of cancer, diabetes, heart, liver, and kidney diseases
* Major gastrointestinal disorders in the past 3 months
* History of heart attacks or stroke
* Unable to meet in-person visit requirements for dining, picking up meals, and tests
* Any mental health condition affecting the ability to provide written informed consent
* If they had not had a routine health checkup 12 months before recruitment.
* If they were unwilling to abstain from taking nutritional supplements, alcohol, non-study foods, and beverages during the study period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
Concentration of phosphatidylcholine in blood | 8 weeks
  Using Microplate Assay

CONTACTS AND LOCATIONS:
Overall Officials: Moul Dey, Ph.D, Principal Investigator — South Dakota State University
Locations (1):
- South Dakota State University, Wagner Hall 416, Brookings, South Dakota, United States

REFERENCES:
- [Derived] Vaezi S, de Vargas BO, Weidauer L, Freeling JL, Dey M. Effects of Minimally Processed Red Meat within a Plant-Forward Diet on Biomarkers of Physical and Cognitive Aging: A Randomized Controlled Crossover Feeding Trial. Curr Dev Nutr. 2025 Dec 10;10(1):107615. doi: 10.1016/j.cdnut.2025.107615. eCollection 2026 Jan. PMID 41551721
- [Derived] Vaezi S, de Vargas BO, Freeling JL, Weidauer L, Dey M. Effects of Minimally Processed Red Meat Within a Plant-Forward Diet on Biomarkers of Physical and Cognitive Aging: A Randomized Controlled Crossover Feeding Trial. medRxiv [Preprint]. 2025 Aug 13:2025.08.11.25333443. doi: 10.1101/2025.08.11.25333443. PMID 40832369